CLINICAL TRIAL: NCT00585260
Title: Mannitol Bronchoprovocation Challenge Ancillary Study Protocol to Best Adjustment Strategy for Asthma Over Long Term
Brief Title: Mannitol Bronchoprovocation Challenge Ancillary Study/ACRN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Syntara (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2007-0071; 144QK18
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Asthma
Keywords: asthma; bronchoprovocation challenge test; mannitol; methacholine
MeSH Terms: conditions — Asthma | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exploratory Mannitol (Experimental): This is an exploratory / ancillary study open to all participants in the BASALT trial [NCT00495157] who consented to undergo mannitol bronchoprovocation procedures during the 36 week treatment period
  Interventions: Drug: mannitol

INTERVENTIONS:
Drug: mannitol — indirect mannitol challenge

SUMMARY:
This is an ancillary study conducted as part of the BASALT trial [NCT00495157].

The overall hypotheses are: 1) an indirect airway challenge procedure using mannitol can safely characterize asthma phenotypes, predict asthma control and exacerbations, predict responses to interventions, and perform more specifically than a direct methacholine challenge and; 2) PX27 pore function in whole blood correlates with measures of airway hyperresponsiveness induced by methacholine and/or mannitol challenges

ELIGIBILITY:
Inclusion Criteria:

* all subjects randomized to the BASALT protocol

Exclusion Criteria:

* positive urine pregnancy test
* requirement for more than two albuterol treatments for reversal of the methacholine bronchoprovocation challenge procedure at visit 4 in the BASALT parent trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02-16 (Actual); Study Completion 2010-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | At 6 weeks, 20 weeks, and 32 weeks
  Mannitol bronchoprovocation challenge testing is safe, effective and well tolerated as compared to methacholine (conducted as part of the main BASALT trial).

OTHER OUTCOMES:
Correlation of the baseline PD15FEV1 with other baseline physiologic measurements collected in the BASALT trial | Baseline
  To evaluate the applicability of mannitol bronchoprovocation to characterize the asthma phenotype. Correlation of the baseline PD15FEV1 with other baseline physiologic measurements and methacholine bronchoprovocation performance as collected in the BASALT trial.

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Sorkness, Pharm.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison Department of Asthma, Allergy and Pulmonary Clinical Research, Madison, Wisconsin, United States

REFERENCES:
- [Background] Calhoun WJ, Ameredes BT, King TS, Icitovic N, Bleecker ER, Castro M, Cherniack RM, Chinchilli VM, Craig T, Denlinger L, DiMango EA, Engle LL, Fahy JV, Grant JA, Israel E, Jarjour N, Kazani SD, Kraft M, Kunselman SJ, Lazarus SC, Lemanske RF, Lugogo N, Martin RJ, Meyers DA, Moore WC, Pascual R, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Boushey HA; Asthma Clinical Research Network of the National Heart, Lung, and Blood Institute. Comparison of physician-, biomarker-, and symptom-based strategies for adjustment of inhaled corticosteroid therapy in adults with asthma: the BASALT randomized controlled trial. JAMA. 2012 Sep 12;308(10):987-97. doi: 10.1001/2012.jama.10893. PMID 22968888